CLINICAL TRIAL: NCT04689620
Title: Helium Neon Laser Versus Gallium Arsenide Laser In Healing Of Venous Ulcers
Brief Title: Helium Neon Laser Versus Gallium Arsenide Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Awad Ramadan Elkholy (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Awad Ramadan Elkholy, principal investigator, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Beni Suef University
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- HELIUM NEON LASER plus regular ulcer care (Experimental): laser scanning the wound with 9.6 jole/cm2 then regular dressing
  Interventions: Device: laser
- GALLIUM ARSENIDE plus regular ulcer care (Experimental): laser scanning the wound with 9.6 jole/cm2 then regular dressing
  Interventions: Device: laser
- regular ulcer care (Active Comparator): dressing for the ulcer
  Interventions: Device: laser

INTERVENTIONS:
Device: laser — treating the venous ulcer with laser

SUMMARY:
There will be different effects for different laser wavelengths in treatment of venous ulcer.

DETAILED DESCRIPTION:
The cost of treating venous ulcer can vary within wide limits and depends on the technology used. In the countries of the European community, the closure of one ulcer as an outpatient procedure costs 800-1500 euros, and supporting anti-relapse treatment makes 100-150 euros per month. In the United States, for closure of venous ulcer within 3 months, direct medical costs reach US$1500- 2000. Prolongation of the treatment for a longer time results in increased cost up to US$30 000 or more.

Poor efficiency of the known methods of treating patients with venous ulcer necessitates the search for new ways and modes of laser therapy (LT) based on a comprehensive approach. Application of physical therapy, primarily with the use of LLLT, capable of influencing various stages in the pathogenesis of the disease, allows a high therapeutic effect in many cases, while ensuring systemic response of the patient's body with the proper exposure procedure.

So, the current study will be conducted to compare the effect of different laser wavelengths on venous ulcers and provide an effective treatment method for patients with venous ulcers with low cost and in short duration.

ELIGIBILITY:
Inclusion Criteria:

* All patients approximately the same age (50-60).
* All patients had venous leg ulcers just above medial malleolus. The common cause of ulcers for all cases was venous insufficiency.
* All patients with conscious.

Exclusion Criteria:

* All patients had no diabetes or blood problems.
* any immunity disorder affect wound heaing.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-26 (Estimated); Primary Completion 2020-12-28 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
wound surface area | two months
  measuring the ulcer surface area by smart phone application
number of bacteria in wound | two months
  measuring number of bacteria by colony count

IPD SHARING:
Plan to Share IPD: Undecided
statistical analysis plan